CLINICAL TRIAL: NCT04274582
Title: The Influences of Chokeberry Extract Supplementation on Redox Status and Body Composition in Handball Players During Competition Phase
Brief Title: The Influences of Chokeberry Extract Supplementation on Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kragujevac (Other)
Responsible Party: Principal Investigator, Isidora Milosavljevic, Assistant professor, University of Kragujevac
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Alixir400protectSportsmen
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Handball Players
Keywords: oxidative stress; handball players; lipid profile; aronia; body composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chokeberry extract consumption (Experimental): The players received 30 mL of liquid chokeberry extract, in the morning before training, once per day for 12 weeks.
  Interventions: Dietary Supplement: chokeberry extract

INTERVENTIONS:
Dietary Supplement: chokeberry extract — The players received 30 mL of liquid chokeberry extract, in the morning before training, once per day for 12 weeks.
  Other Names: Alixir400protect

SUMMARY:
The study included 16 handball players, aged 16-24 years , of handball club "Novi Beograd". All study participants were apparently healthy, had no active sports injuries, did not use any medications, and were non-smokers. Standardized questionnaires conducted under the supervision of a trained nutritionist were used to collect general data, nutritional habits and use of dietary supplements. The athletes who used any dietary supplements at least a month before the study, were excluded. All participants (or their parents if they were under the age of 18) signed an informed consent document. The study was approved by the Ethical committee of The Military Medical Academy, Belgrade.

The study was conducted during regular competition season, and lasted for twelve weeks. All participants had the same training and nutritional regime, which excluded intake of berries. The players received 30 mL of liquid chokeberry extract, in the morning before training, once per day for 12 weeks. For the preparation of chokeberry extract (liquid form) was used fruit (berries) of Aronia melanocarpa Elliot, Rosaceae. The extract was donated by Pharmanova Belgrade, Serbia. Process of extraction is performed under specific conditions which are subject of technical patent (producer EUHEM), for the purpose of production of extract with high concentration of polyphenols. The design of the product included few demands: sufficient daily dose of polyphenols to be dietary supplement, small volume which can be consumed as shot and acceptable taste for most consumers. Compliance was monitored by the trainers.

ELIGIBILITY:
Inclusion Criteria:

* healthy handball players of handball club "Novi Beograd" during competition phase.

Exclusion Criteria:

* active sports injuries,
* usage of any medications,
* smokers

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — In study the male handball players were onlz included.
Enrollment: 16 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Superoxide anion radical | three months
  The concentration of O2- was measured after the reaction of nitro blue tetrazolium in TRIS buffer with plasma at 530 nm.
hydrogen peroxide | three months
  The determination of H2O2 concentration is based on oxidation of phenol red using hydrogen peroxide, in reaction catalyzed by enzyme peroxidase from horse radish (POD). The level of H2O2 was measured at 610 nm.
nitrites | three months
  Nitric oxide (•NO) decomposes rapidly to form stable metabolite nitrite/nitrate products. The method for detection of the plasma nitrite levels is based on the Griess reaction. Nitrites (NO2-) were determined as an index of NO production with Griess reagent (forms purple diazocomplex). Nitrites were measured at 550 nm.
index of lipid peroxidation | three months
  The degree of lipid peroxidation in the plasma was estimated by measuring the TBARS using 1% thiobarbituric acid in 0.05 NaOH, incubated with plasma at 100 C for 15 min, and measured at 530 nm.

SECONDARY OUTCOMES:
Superoxide dismutase | three months
  SOD activity was determined by the epinephrine method of Beutler. 100 μl lysate and 1 mL of carbonate buffer were mixed; then 100 μl of epinephrine was added. Detection was performed at 470 nm.
Reduced glutathione | three months
  The level of GSH was determined based on GSH oxidation with 5.5- dithio-bis-6.2-nitrobenzoic acid using the method reported by Beutler.
Catalase | three months
  CAT activity was determined according to Aebi. Lysates were diluted with distilled water (1:7 v/v) and treated with chloroform-ethanol (0.6:1 v/v) to remove haemoglobin; then 50 ll of CAT buffer, 100 μl of sample, and 1 mL of 10 mM H2O2 were added to the samples. Detection was performed at 360 nm.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medical Science, Kragujevac, Serbia

IPD SHARING:
Plan to Share IPD: No